CLINICAL TRIAL: NCT00362973
Title: Early Assessment of Response to Targeted Breast Cancer Therapy
Brief Title: PET Scans in Assessing Response To Treatment in Patients Receiving Hormone Therapy or Trastuzumab for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Hannah Linden, MD, FHCRC
Other Study IDs: 6213; P30CA015704 (NIH); UWCC-6213; UWCC-06-0445-H/D; CDR0000492255 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Biopsy, Needle; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Hormone Receptor Positive Breast Cancer: Patients with hormone receptor positive primary, recurrent or metastatic breast cancer with a treatment plan that involves (neoadjuvant) administration of aromatase inhibitor and ovarian suppression (if premenopausal).
  Interventions: Other: laboratory biomarker analysis; Procedure: needle biopsy; Procedure: positron emission tomography; Procedure: radionuclide imaging; Radiation: fludeoxyglucose F 18
- HER-2/neu Positive Breast Cancer: Patients with HER-2/neu positive primary, recurrent or metastatic breast cancer with a treatment plan that involves (neoadjuvant) administration of trastuzumab.
  Interventions: Other: laboratory biomarker analysis; Procedure: needle biopsy; Procedure: positron emission tomography; Procedure: radionuclide imaging; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Other: laboratory biomarker analysis
Procedure: needle biopsy
Procedure: positron emission tomography
Procedure: radionuclide imaging
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic procedures, such as PET scans, may help in learning how well hormone therapy and trastuzumab work to kill breast cancer cells and allow doctors to plan better treatment.

PURPOSE: This clinical trial is studying how well PET scans work in assessing response to treatment in patients receiving hormone therapy or trastuzumab for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate the percent change in fludeoxyglucose F 18 (FDG)-positron emission tomography (PET) standardized uptake value (SUV) and percent change in cell proliferation (as assessed by tumor biopsy) during hormonal therapy with tumor response in patients with hormone receptor-positive (estrogen receptor or progesterone receptor) breast cancer.
* Correlate the percent change in FDG-PET SUV and percent change in cell proliferation (as assessed by tumor biopsy) during treatment with trastuzumab (Herceptin®) with tumor response in patients with HER-2/neu-positive breast cancer.
* Compare the association between two-week changes in cell proliferation rate (as measured by FDG-PET and biopsy) in patients treated with an aromatase inhibitor or trastuzumab.

OUTLINE: Patients are assigned to 1 of 2 groups according to therapy.

* Group 1 (patients receiving hormonal therapy): Patients undergo fludeoxyglucose F 18-positron emission tomography (FDG-PET) scan and may also undergo 16α-fluoroestradiol F 18 (FES)-PET scan at baseline (prior to beginning therapy) and FDG-PET scan 2 weeks after beginning therapy.

Blood samples are collected at baseline and at 3 and 6 months after beginning aromatase inhibitor therapy. The blood samples are examined for hormone levels, including estradiol, estrone, testosterone, follicle-stimulating hormone, and sex hormone-binding globulin.

* Group 2 (patients receiving HER-2/neu targeted therapy): Patients undergo biopsy and FDG-PET scan at baseline (prior to beginning therapy) and FDG-PET scan 1-2 weeks after beginning therapy.

Some patients undergo a core-needle biopsy 2 weeks after beginning therapy. Biopsies are assessed for the following markers: proliferative rate (Ki67), estrogen receptor, progesterone receptor, HER-2/neu, epidermal growth factor receptor, androgen receptor, and topoisomerase II.

After completion of study therapy, patients are followed periodically for 6 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed breast cancer with 1 of the following:

  * Hormone receptor-positive disease and planning to receive treatment with neoadjuvant aromatase inhibitor and ovarian suppression therapy (if premenopausal)
  * Recurrent and/or metastatic hormone receptor-positive disease and planning to receive treatment with an aromatase inhibitor and ovarian suppression therapy (if premenopausal)
  * Metastatic HER-2/neu-positive disease and planning to receive treatment with neoadjuvant trastuzumab (Herceptin®)
  * Recurrent HER-2/neu-positive disease and planning to receive treatment with trastuzumab (Herceptin®)
* Tumor must be accessible for biopsy and assessable for response

  * Tissue block must be available for review of experimental markers or patient must be willing to undergo biopsy
* Evaluable disease by FDG-PET scan
* Available for positron emission tomography (PET) imaging with a clinical indication for PET scan

  * May aslo be enrolled on an experimental nuclear imaging study of 16α-fluoroestradiol F 18-PET scan (if hormone positive)
* Concurrently receiving treatment (hormonal or other) for breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

* Female or male
* Postmenopausal or premenopausal
* Life expectancy ≥ 2 months
* No uncontrolled diabetes mellitus or other comorbidity that would preclude imaging
* Not pregnant
* Negative pregnancy test
* Able to tolerate scanning (e.g., no claustrophobia or severe pain)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent participation on another clinical study or other imaging studies allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary, recurrent or metastatic breast cancer that is either hormonal receptor positive or HER-2/neu positive.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2006-05; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Percent change in fludeoxyglucose F 18-positron emission tomography (FDG-PET) standardized uptake value and change in markers of proliferation (Ki67) at 2 weeks | 2 weeks
Percent change in cell proliferation correlated with absolute measures of FDG-PET | 2 weeks
Correlation of early FDG-PET with response prediction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hannah M. Linden, MD, Principal Investigator — Seattle Cancer Care Alliance
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington